CLINICAL TRIAL: NCT06964984
Title: Effects of Virtual Glasses, Stress Ball and Music Intervention on Pain, Anxiety and Comfort in Patients Undergoing Inguinal Hernia Surgery: A Randomized Controlled Trial
Brief Title: Effects of Virtual Glasses, Stress Ball and Music Intervention on Pain, Anxiety and Comfort in Patients Undergoing Inguinal Hernia Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cagla Toprak (Other)
Responsible Party: Sponsor-Investigator, Cagla Toprak, Dr., Atlas University
Organization: Atlas University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23.12.2024- 10/40
Record Dates: First submitted 2025-04-04; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Pain; Anxiety; Inguinal Hernia
Keywords: inguinal hernia,virtual reality,stress ball,music therapy
MeSH Terms: conditions — Pain; Anxiety Disorders; Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- music group (Experimental): The patient will be asked to choose their favorite music. The playlist will include ten songs from each music group (pop, Turkish classical music, local folk songs and religious music), for a total of 50 songs. The options will be shown to the patient via the phone (Apple/ MU783TU/A) and the music they want will be added to the playlist. The selected music will be listened to for 15 minutes before the surgery.
  Interventions: Other: Music intervention; Other: stres ball; Other: Virtual Reality Glasses
- stress ball (Experimental): Stress balls will be given to the patient in both palms, and they will be asked to count from one to five and squeeze them twice. The patient will be shown how to use the stress balls for 15 minutes before the surgery and will be made to practice. When the 15 minutes are up, the nurse will inform the patient and have the patient put the balls down.
  Interventions: Other: Music intervention; Other: stres ball; Other: Virtual Reality Glasses
- virtual reality glasses (Experimental): The patient will be shown a video of a nature walk by the nurse providing nursing care to the patient. The patients will be shown a video with virtual reality glasses for 15 minutes before the surgery.
  Interventions: Other: Music intervention; Other: stres ball; Other: Virtual Reality Glasses
- control group (No Intervention): Patients in the control group will not undergo any intervention other than the standard care protocol.

INTERVENTIONS:
Other: Music intervention — The patient will be asked to choose their favorite music. The playlist will include ten songs from each music group (pop, Turkish classical music, local folk songs and religious music), a total of 50 songs. The options will be shown to the patient via the phone (Apple/ MU783TU/A) and the music they want will be added to the playlist. The selected music will be listened to for 15 minutes before the surgery.
  Arms: music group; stress ball; virtual reality glasses
Other: stres ball — Stress balls will be given to the patient in both palms, they will be asked to count from one to five and squeeze twice. The patient will be shown and made to use the stress balls for 15 minutes before the surgery. When the 15 minutes are up, the patient will be informed by the nurse and the patient will be asked to release the balls.
  Arms: music group; stress ball; virtual reality glasses
Other: Virtual Reality Glasses — The patient will be shown a video of a nature walk by the nurse providing nursing care to the patient. The patients will be shown a video with virtual reality glasses for 15 minutes before the surgery.
  Arms: music group; stress ball; virtual reality glasses

SUMMARY:
Although it changes with age, due to its high incidence and prevalence, inguinal hernia is one of the most commonly performed surgeries by general surgeons. Pain, anxiety and changes in comfort levels in patients after inguinal hernia repair surgery negatively affect the patient's recovery after surgery. One of the goals of nursing care practices in the perioperative period, especially in patients undergoing surgery, is to provide and maintain patient comfort. Today, the concept of comfort is a part of quality nursing care, allowing patients to be comfortable, carefree, recover more quickly and cope better with disease stress. Using non-pharmacological methods in pain management reduces the use of pharmacological methods, increases the patient's comfort level, reduces stress and anxiety, increases the individual's sense of control over their own health and increases physical function and daily life activities. Virtual reality, music therapy, stress ball are used in various areas of clinical medical care as a way to distract attention and relieve pain.

DETAILED DESCRIPTION:
This study aimed to evaluate the effects of distraction methods such as virtual reality, music therapy and stress ball applications on pain, anxiety and comfort levels in patients undergoing inguinal hernia surgery.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-70 Inguinal surgery will be performed,

  * No communication problems, can speak Turkish,
  * No psychiatric illness or mental perception problems,
  * No vision, hearing and perception problems,
  * No physical problems in squeezing a stress ball,

Exclusion Criteria:

* • Any postoperative complications,

  * Patients who do not agree to participate in the study,
  * Patients using anxiolytic drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-05 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
comfort | 10 minutes before surgery stress.
  t was designed by researchers similar to the use of "Visual Analog Scale (VAS)". VAS is used to make measurable some values that cannot be measured numerically, which are evaluated by individuals by marking on a horizontal or vertical line of 10 cm or 100 mm, one end of which indicates that the individual is "very good" and the other end indicates that the individual is "very bad".
pain assessment | 10 minutes before surgery pain
  It was designed by researchers similar to the use of "Visual Analog Scale (VAS)". VAS is used to make measurable some values that cannot be measured numerically, which are evaluated by individuals by marking on a horizontal or vertical line of 10 cm or 100 mm, one end of which indicates that the individual is "very good" and the other end indicates that the individual is "very bad".
anxiety | 10 minutes after surgery
  This scale consists of two parts: STAI-I and STAI-II. The scale consists of 20 items. Items 1-20 on the scale measure anxiety in four options. Trait anxiety scores were calculated by adding the unchanging number 35 for the trait anxiety scale to the obtained result. The lowest score on the scale is 20, the highest score is 80. Score Status Anxiety level; 0-19 points indicate no anxiety, 20-39 points indicate mild anxiety, 40-59 points indicate moderate anxiety, 60-79 points indicate severe anxiety, 80 and above indicate panic level anxiety. As the score increases, the anxiety level also increases.
comfort | Will be evaluated at 10 minutes and 24 hours after surgery
  It was designed by researchers similar to the use of "Visual Analog Scale (VAS)". VAS is used to make measurable some values that cannot be measured numerically, which are evaluated by individuals by marking on a horizontal or vertical line of 10 cm or 100 mm, one end of which indicates that the individual is "very good" and the other end indicates that the individual is "very bad".
pain assesment | Will be evaluated at 10 minutes and 24 hours after surgery
  It was designed by researchers similar to the use of "Visual Analog Scale (VAS)". VAS is used to make measurable some values that cannot be measured numerically, which are evaluated by individuals by marking on a horizontal or vertical line of 10 cm or 100 mm, one end of which indicates that the individual is "very good" and the other end indicates that the individual is "very bad".
anxiety | Will be evaluated at 10 minutes and 24 hours after surgery
  this scale consists of two parts: STAI-I and STAI-II. The scale consists of 20 items. Items 1-20 on the scale measure anxiety in four options. Trait anxiety scores were calculated by adding the unchanging number 35 for the trait anxiety scale to the obtained result. The lowest score on the scale is 20, the highest score is 80. Score Status Anxiety level; 0-19 points indicate no anxiety, 20-39 points indicate mild anxiety, 40-59 points indicate moderate anxiety, 60-79 points indicate severe anxiety, 80 and above indicate panic level anxiety. As the score increases, the anxiety level also increases.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Dogan Yilmaz E, Unlusoy Dincer N. The Effects of Virtual Reality Glasses on Vital Signs and Anxiety in Patients Undergoing Colonoscopy: A Randomized Controlled Trial. Gastroenterol Nurs. 2023 Jul-Aug 01;46(4):318-328. doi: 10.1097/SGA.0000000000000733. Epub 2023 Jun 5. PMID 37278621
- See also: The Effect of Virtual Reality on Pain and Anxiety During Colonoscopy: A Randomized Controlled Trial — https://pubmed.ncbi.nlm.nih.gov/34231475/
- See also: The Effect of Virtual Reality on Pain Experienced by School-Age Children During Venipuncture: A Randomized Controlled Study — https://pubmed.ncbi.nlm.nih.gov/37466456/
- See also: Use of virtual reality in managing paediatric procedural pain and anxiety: An integrative literature review — https://pubmed.ncbi.nlm.nih.gov/35068011/